CLINICAL TRIAL: NCT05214209
Title: Addressing Disparity in Diabetes Prevention Through Digital Health Supported PRe-diabetes Intervention, Management and Evaluation (PRIME) Program Based in Malaysian Community Pharmacies: A Pilot Study
Brief Title: Diabetes Prevention and Prediabetes Management in Adult
Acronym: PRIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University (Other)
Collaborators: Caring Pharmacy (Unknown); Bionime Corporation (Industry)
Responsible Party: Principal Investigator, Shaun Lee Wen Huey, Associate Professor, Monash University Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRIME (pilot)
Record Dates: First submitted 2021-12-15; First posted 2022-01-28 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: PreDiabetes
Keywords: Digital Health; Mobile Health; Lifestyle Program; Prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Cluster randomisation with blinding of statisticians
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): Participants receiving the phone app together with a fitness tracker. All participants will receive the educational curriculum over a period of 4 weeks through the app. The mobile app allows secure patient monitoring through a participant dashboard that the coach can use to increase patient adherence and motivation to achieve goals. The participant can use the app to log their food intake, weight, steps, exercise, in addition to participating in the peer support via the chat function. Participants will also receive regular care and follow up in community pharmacies for support.
  Interventions: Behavioral: Digital health supported
- Usual care arm (Active Comparator): The control group will be a "usual care" condition in which participants are free to seek any assistance for their medical care during the study period. Participants will be given physical tracking sheets to record their food intake, weight, steps and exercises.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Digital health supported — Participants will be issued a fitness tracker, a Bluetooth enabled glucometer, and a custom developed app which they can communicate digitally to the study investigators either as a group or individually. In the beginning of the study, participants will be taught on how to use the program, how to interact with their coach, and the importance of maintaining motivation throughout the program. Participants will have access to a pharmacist-participant messaging, group messaging, daily challenges for behavior change, education articles (weekly bite-sized content over 4 weeks), food logging, steps and exercise logging, and feedback. They will be asked to log their weight, meals, and physical activity within the program on a weekly basis. Pharmacist will monitor participant progress through a web-based dashboard. Community pharmacist will be assisting users in setting specific, measurable, attainable, realistic, and time-based goals on a weekly basis.
  Arms: Intervention arm
Behavioral: Usual care — Participants will be issued a fitness tracker and Bluetooth enabled glucometer but these functions will not be enabled or linked to any app. All participants will be given physical tracking sheets to log in their food intake, blood glucose levels and food diary but will not have access to a personal coaching. Participants are free to seek any assistance for their medical care during the study period.
  Arms: Usual care arm

SUMMARY:
Currently, an estimated 3.9 million Malaysians continue to live with diabetes with many more who live with prediabetes. Diabetes was the one of the leading causes of death in the Malaysia and the leading cause for kidney failure, lower-limb amputations, and adult-onset blindness. Heart disease and stroke are two to four times more likely for individuals with diabetes. The use of mHealth or mobile health application can reduce blood sugar among individuals with prediabetes but also prevent a later occurrence of diabetes. In this study, the investigators aim to develop and evaluate the effectiveness of a digital health supported pre-diabetes management program based in an urban community pharmacy setting

DETAILED DESCRIPTION:
Pre-diabetes is an intermediate state of hyperglycaemia with glycaemic parameters above normal but below the type 2 diabetes mellitus (T2DM) threshold. It was estimated that >25% of individuals who are pre-diabetic convert to T2DM within 3-5 years and 70% of individuals with pre-diabetes will develop into full-fledge T2DM within their lifetimes. According to the 2017 estimate, the disease burden of pre-diabetes at Western Pacific region was 7.6% (126.7 millions). The situation is more alarming in Malaysia where a national pre-diabetes prevalence of 22.1% was noted. Currently available support and self-care services offered in Public Hospitals such as the Diabetes Mellitus Treatment Adherence Clinics (DMTAC) are managed based on the in-person appointment basis. Most of the clinics are available only in specific locations. The need to travel long distance as well as long waiting hours has deterred the success of the programs. This is particularly true for the urban poor who are less likely to take time off from work than those from the higher income group. It is also noteworthy to state that the management program when available, generally target the diagnosed T2DM patients.

Studies have shown that individuals with pre-diabetes can substantially reduce their risk of progression to T2DM via participation in evidence-based lifestyle change programs. Previous reports have recorded 54-58% reduction in risk for development to T2DM over 1-3 years with the protective benefit persisting up to 10 years following completion of the program. However, there are several considerations when implementing effective lifestyle intervention program among the pre-diabetes populations in Malaysia. The intervention program should easily be accessible and not confined to public primary and secondary healthcare centres which are already suffering from an overcapacity. Furthermore, consultation should be provided by properly trained healthcare professionals while the ease of communication between the patients and the "lifestyle coach" should be made available.

The advancement of information technology coupled with the increasing availability and acceptance of internet and mobile devices provide useful opportunities for application of wireless and mobile technology in order to enhance self-management of chronic conditions. The incorporation of digital technologies can improve patient adherence and facilitate real-time monitoring of vital biological measurements (i.e. via wearable). Additionally, the "mobile health" (mHealth) services are easily scalable, thus providing opportunities to a greater public accessibility and narrow the disparity in access to disease management. In this study, the investigators propose to pilot a digital health supported pre-diabetes management program based in an urban community pharmacy setting

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above
* BMI 23 and above
* HbA1c 5.7 - 6.3%

Exclusion Criteria:

* Unable to give informed consent
* Pregnant or lactating
* Established diabetes
* Terminal illness
* Does not own a mobile phone
* Plans to relocate to an area or travel plans that do not permit full participation in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of mobile app assessed by the engagement rate with the mobile app | 1 month
  Engagement rate with the mobile app will be measured via time spend on using the app functions, measured in hours.
Acceptability of mobile app assessed by a semi-structured interview | 1 month
  Semi-structured interview focusing on users experience will be conducted post-intervention.

SECONDARY OUTCOMES:
Change in health related quality of life as accessed by EuroQol (EQ-5D-5L) | Baseline, 1 month
  The questionnaire assess patient's health state in 5 dimensions- anxiety/depression, mobility, self-care, usual activities, pain/discomfort. Each dimension can be scored from 1 - 5, summing up to a total score of between 5 - 25. A lower score representing a better health state.
Change in dietary practice | Baseline, 1 month
  3-Day diet recall to assess changes in food intake
Change in physical activity | Baseline, 1 month
  Physical Activity Questionnaire (short form) (IPAQ) to obtain internationally comparable data on health-related physical activity. Time spent on physical activities will be measured and converted into metabolic equivalent for task (MET). A lower MET indicates a lower physical activity level.
Change in blood pressure | Baseline, 1 month
  Systolic and diastolic pressures will be collected during the study period, unit in mmHg
Change in lipid profile | Baseline, 1 month
  HDL, LDL, triglycerides and total cholesterol levels will be collected, unit in mmol/L
Change in knowledge, attitude and practice towards prediabetes | Baseline, 1 month
  Knowledge Attitude Practice-Prediabetes Assessment Questionnaire (KAP-PAQ) questionnaire will be administered pre- and post intervention. The minimum total score is 14 while the maximum total score is 91. A higher score indicating a better knowledge, attitude and practice.
Change in weight | Baseline, 1 month
  Weight Loss by % of change and total weight change (kg).
Change in body fat composition | Baseline, 1 month
  Body fat composition change measured in % change.
Change in waist-to-hip ratio | Baseline, 1 month
  Waist circumference and hip circumference measured in centimetres.

CONTACTS AND LOCATIONS:
Overall Officials: Shaun Lee, PhD, Principal Investigator — Monash University Malaysia; Chun Wie Chong, PhD, Principal Investigator — Monash University Malaysia
Locations (1):
- School of Pharmacy, Subang Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share any related individual participant data within reasonable request which can be obtained from the principal investigators